CLINICAL TRIAL: NCT02182180
Title: Surgical Critical Care InitiativeTissue and Data Acquisition Protocol
Brief Title: SC2i Tissue and Data Repository Protocol
Acronym: SC2i
Status: Recruiting | Type: Observational
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency); United States Department of Defense (U.S. Federal Agency); Duke University (Other); Emory University (Other); Grady Health System (Other); Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: SC2I SUR902506; HT94041310032 (Other: HJF/USUHS)
Record Dates: First submitted 2014-06-27; First posted 2014-07-08 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Protocol participants: All participants enrolled on the protocol

SUMMARY:
The purpose of this study is to collect samples of blood, urine, cerebrospinal fluid (CSF, the fluid that surrounds the brain and spinal cord), wound tissue and/or wound fluids, and other body fluids and tissues from people who have been seriously injured or ill. The samples will be used to develop and assess tests and/or tools that doctors can use to decide the best treatment plan for seriously injured or ill military personnel and for civilians. Additonal protocols to use the samples will be submitted as separate protocols.

ELIGIBILITY:
Inclusion Criteria:

* Patients with injury or illness requiring surgical care or treatment in a critical care or emergency setting who are being cared for at SC2I sites (Grady Memorial Hospital, Emory Univeristy Hospital, and Duke University Health Systems)
* Healthy volunteer control subjects to include individuals without any known injury or end-stage organ disease and patients who have recovered from prior injury.
* Ability to understand the purposes and risks of the study and willingly give written informed consent, or in the case of incapacitated patients, a willing surrogate able to give written informed consent.

Exclusion Criteria:

* Any condition that, in the opinion of the attending physician, would place the patient or volunteer subject at undue risk by participating. Specific conditions include but are not limited to anemia prohibitive of phlebotomy, coagulopathy, or technical considerations that would prevent acquisition of sufficient tissue or fluid for clinical use. Acquisition of samples from patients requiring active transfusion or with transfusion-associated coagulopathy will be considered as appropriate study candidates at the discretion of the attending physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with injury or illness requiring surgical care or treatment in a critical care or emergency setting who are being cared for at SC2I sites, including Grady Memorial Hospital, Emory University Hospital, and Duke University Health System. Also, healthy volunteer control subjects to include individuals without any known injury or end-stage organ disease and patients who have recovered from prior injury.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2014-09-09 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Collecting, processing and archiving human tissue | Samples will be stored indefinitely in repository
  Samples of blood, urine, cerebrospinal fluid, wound tissue and/or wound fluids, and other body fluids and tissues from people who have been seriously injured or ill will be collected. The samples will be used to develop and assess tests and/or tools that doctors can use to decide the best treatment plan for seriously injured or ill military personnel and for civilians. Additional research on the samples will be under separate protocols. This is a collection protocol.

CONTACTS AND LOCATIONS:
Overall Officials: CAPT Eric Elster, MD, US Navy, Study Director — Uniformed Services University of the Health Sciences; Allan M. Kirk, MD, PhD, Principal Investigator — Duke University; Timothy G Buchman, Ph.D, MD, Principal Investigator — Emory University; Christopher J. Dente, MD, Principal Investigator — Grady Hospital; Benjamin K Potter, MD, FACS, Principal Investigator — Uniformed Services University - Walter Reed Surgery
Locations (4):
- United States (4):
  - Grady Health Systems, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Duke University Health Systems, Durham, North Carolina

REFERENCES:
- [Derived] Haines KL, Li R, Grey S, Kim HE, Gann E, Almond C, Rouse M, Joshi M, Schobel S, Agarwal S, Kirk A, Elster E, Fernandez-Moure JS. Exploratory cluster analysis of IL2Ra and associated biomarkers and complications after blunt chest trauma. J Trauma Acute Care Surg. 2025 Jun 1;98(6):899-906. doi: 10.1097/TA.0000000000004568. Epub 2025 Apr 14. PMID 40223169
- [Derived] Rindler RS, Robertson H, De Yampert L, Khatri V, Texakalidis P, Eshraghi S, Grey S, Schobel S, Elster EA, Boulis N, Grossberg JA. Predicting Vasospasm and Early Mortality in Severe Traumatic Brain Injury: A Model Using Serum Cytokines, Neuronal Proteins, and Clinical Data. Neurosurgery. 2024 Oct 11. doi: 10.1227/neu.0000000000003224. Online ahead of print. PMID 39471078
- [Derived] Gerardo CJ, Silvius E, Schobel S, Eppensteiner JC, McGowan LM, Elster EA, Kirk AD, Limkakeng AT. Association of a Network of Immunologic Response and Clinical Features With the Functional Recovery From Crotalinae Snakebite Envenoming. Front Immunol. 2021 Mar 15;12:628113. doi: 10.3389/fimmu.2021.628113. eCollection 2021. PMID 33790901
- See also: Henry M. Jackson Foundation for the Advancement of Military Medicine, Inc. — http://www.hjf.org
- See also: Uniformed Services University of the Health Sciences — http://www.usuhs.edu
- See also: Grady Health Systems — http://www.gradyhealth.org/
- See also: Duke University Medical Center — http://www.dukemedicine.org/
- See also: Emory Healthcare — http://www.emoryhealthcare.org